CLINICAL TRIAL: NCT07114094
Title: Development and Validation of a Deprescribing Tool Relevant to the Indian Context and Evaluation of Its Effectiveness in Reducing Inappropriate Polypharmacy in the Elderly
Brief Title: Development, Validation and Evaluation of a Deprescribing Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Collaborators: St Johns Medical College Hospital, Bangalore, India (Other)
Responsible Party: Principal Investigator, Ratinder Jhaj, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20032
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Elderly
Keywords: Deprescribing Tool; Polypharmacy; Elderly

STUDY DESIGN:
Intervention Model Description: Cluster Randomized ( Participating Prescribers are randomized, not patients) Open Label, Delayed or Sequential Intervention Trial. Intervention arm will begin after completion of Control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Prescribers in this arm will not use the Deprescribing Tool, and will prescribe as per routine practice.
- Intervention Arm (Experimental): Prescribers in this arm will be trained in the use of the Deprescribing Tool and provided the Tool for medication review during patient consultation. The prescriber will be encouraged to refer to the tool for medication review of elderly patients aged ≥ 60 years and take deprescribing decision if indicated.
  Interventions: Other: Deprescribing Tool

INTERVENTIONS:
Other: Deprescribing Tool — Deprescribing Tool will be used for medication review during patient consultation. The prescriber will be encouraged to refer to the tool for medication review of elderly patients aged ≥ 60 years and take deprescribing decision if indicated.
  Deprescribing may take place in any of the following ways-
  1. Immediate discontinuation of a drug, e.g., a duplicate drug
  2. Initiation of gradual tapering of a drug e.g., an anxiolytic, which is no longer indicated
  3. Reduction in dose of a drug, e.g., lower dose of an NSAID for relief of symptoms of rheumatoid arthritis Only 1-3 medicines will be deprescribed at a time. Medicines with overlapping indications will not be deprescribed at the same time so it is clear which medicine is responsible if withdrawal effects occur.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to learn if a deprescribing tool can help in reducing prescriptions with potentially inappropriate medications (PIMs), in the Indian elderly population. The main question it aims to answer is- Can inappropriate polypharmacy in elderly patients be reduced through development and implementation of a deprescribing tool relevant to the Indian context? Researchers will compare control arm outcome parameters to see if there is a reduction in Proportion of prescriptions with at least one PIM ( Primary outcome parameter).

Participating Prescribers ( Physicians) will be randomized to Control or Intervention arms. Particpating patients will not be randomized, and will receive routine consultation with a Physician who does not use the Deprescribing Tool (Control arm) or a prescriber who uses the Deprescribing tool ( Intervention Arm)

DETAILED DESCRIPTION:
Rationale: Polypharmacy is common in the elderly and is associated with increased risk of serious adverse events, including falls, cognitive impairment, functional decline, hospitalization, and death. In addition, some of the prescribed drugs may be potentially inappropriate medications (PIM), whose risks outweigh their benefits. It is therefore necessary to review medication intake of the elderly and discontinue or reduce the dose of the ones that are no longer required. This process, termed deprescribing, can reduce prescription of PIMs, improving prescription quality and minimize risks due to potential adverse effects and drug-disease or drug-drug interactions, as well as cost of therapy. Novelty: Although there are many tools for deprescribing, none of these tools has been developed for the Indian context, where there is widespread use of fixed dose combinations (FDCs), use of medicines from different systems of medicines, and high out of pocket expenditure on medicines. Also, some of the medications listed in existing tools are not marketed in India, while some which are commonly prescribed in the country are not listed in the tools. We therefore propose to develop and validate a deprescribing tool for the Indian elderly population, evaluate its impact on prescription quality and risk minimization, as well as explore the facilitators and barriers in the implementation of the tool. Study Design: Multicenter multi-method study. Deprescribing tool will be developed through a modified Delphi method. Prescribers will then be enrolled and randomised to either the control or intervention arm. Prescribers in control arm will prescribe as routine practice, without the aid of the tool. Prescribers in the intervention arm will use the deprescribing tool for medication review and deprescription, if indicated. Elderly patients (≥ 60 years old) of either sex, will be identified by research staff at the OPD registration counter, and approached to consent for the study. Prescriptions of consenting patients (≥ 60 years) will be photographed after consultation with prescriber in either arm. Prescriptions from both arms will be compared for assessment of outcome parameters. Sample size: 1650 (825 per study site) patients will be included evaluation of effectiveness of the tool. To evaluate barriers and facilitators to implementation, in depth interviews will be held with all 30 prescribers (15 at each site). Follow-up: Patients will be followed up at one month telephonically (or in person in case of a routine follow up visit at one month) to inquire about any adverse events, including hospitalization due to any cause. Patients will also be provided with the contact number of a study staff to be contacted in case of any problem within or after the one month follow up period. Expected Outcome: Improved quality of prescribing in the elderly, with reduction in proportion of prescriptions with PIMs, reduction in average number of PIMs prescribed per prescription and reduction of ADRs, drug-disease and drug-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (≥ 60 years) of either sex, visiting the General Medicine/ Community and Family Medicine OPD of the study sites

Exclusion Criteria:

* Patients not willing to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Proportion of prescriptions with at least one PIM | From enrollment to end of consultation at 30 minutes to 1 hour
  Proportion of prescriptions with at least one PIM in the control arm minus proportion of prescriptions with at least one PIM in the intervention arm.
  Proportion= Number of prescriptions with at least one PIM ÷Total number of prescriptions included in the respective arm (intervention/control)

SECONDARY OUTCOMES:
Change in Average number of PIMs per prescription | From enrollment to the end of consultation at 30 minutes to 1 hour
  Average number of PIMs in control arm minus Average number of PIMs in intervention arm
  Average = Number of PIMs ÷ Total number of prescriptions included in the respective arm (intervention/control)
Change in Proportion of prescriptions in which at least one PIM was deprescribed | From enrollment to the end of consultation at 30 minutes to 1 hour
  Proportion of prescriptions in which at least one PIM was deprescribed in the intervention arm minus Proportion of prescriptions in which at least one PIM was deprescribed in the control arm
  Proportion=Number of prescriptions in which at least one PIM was deprescribed ÷Total number of prescriptions included in the respective arm (intervention/control)
Change in Average number of Potential ADRs, Drug- Drug Interactions and Drug- Disease Interactions | From enrollment to the end of consultation at 30 minutes to 1 hour
  Average number of Potential ADRs, Drug- Drug Interactions and Drug- Disease Interactions in the control arm minus Average number of Potential ADRs, Drug- Drug Interactions and Drug- Disease Interactions in the intervention arm
  Average: Number of Potential ADRs, Drug- Drug Interactions and Drug- Disease Interactions ÷ Total number of patients in the respective arm (intervention/control)
Change in Average number of Adverse Events at one month | 1 month
  Average number of Adverse Events in the control arm minus Average number of Adverse Events in the intervention arm Average: Number of Adverse Events÷ Total number of patients in the respective arm (intervention/control)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jerin J Cherian, MD, Study Chair — Indian Council of Medical Research and Karolinska Institute, Sweden
Locations (2):
- India (2):
  - St. John's Medical College, Bangalore, India, Bangalore, Karnataka
  - All India Institute of Medical Sciences Bhopal, Bhopal, Madhya Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Candeias C, Gama J, Rodrigues M, Falcao A, Alves G. Potentially Inappropriate Medications and Potential Prescribing Omissions in Elderly Patients Receiving Post-Acute and Long-Term Care: Application of Screening Tool of Older People's Prescriptions/Screening Tool to Alert to Right Treatment Criteria. Front Pharmacol. 2021 Oct 19;12:747523. doi: 10.3389/fphar.2021.747523. eCollection 2021. PMID 34737705
- [Background] By the 2023 American Geriatrics Society Beers Criteria(R) Update Expert Panel. American Geriatrics Society 2023 updated AGS Beers Criteria(R) for potentially inappropriate medication use in older adults. J Am Geriatr Soc. 2023 Jul;71(7):2052-2081. doi: 10.1111/jgs.18372. Epub 2023 May 4. PMID 37139824
- [Background] Bhagavathula AS, Vidyasagar K, Chhabra M, Rashid M, Sharma R, Bandari DK, Fialova D. Prevalence of Polypharmacy, Hyperpolypharmacy and Potentially Inappropriate Medication Use in Older Adults in India: A Systematic Review and Meta-Analysis. Front Pharmacol. 2021 May 19;12:685518. doi: 10.3389/fphar.2021.685518. eCollection 2021. PMID 34093207
- [Background] O'Mahony D, Cherubini A, Guiteras AR, Denkinger M, Beuscart JB, Onder G, Gudmundsson A, Cruz-Jentoft AJ, Knol W, Bahat G, van der Velde N, Petrovic M, Curtin D. STOPP/START criteria for potentially inappropriate prescribing in older people: version 3. Eur Geriatr Med. 2023 Aug;14(4):625-632. doi: 10.1007/s41999-023-00777-y. Epub 2023 May 31. PMID 37256475
- [Background] Renom-Guiteras A, Meyer G, Thurmann PA. The EU(7)-PIM list: a list of potentially inappropriate medications for older people consented by experts from seven European countries. Eur J Clin Pharmacol. 2015 Jul;71(7):861-75. doi: 10.1007/s00228-015-1860-9. Epub 2015 May 14. PMID 25967540
- [Background] Ibrahim K, Cox NJ, Stevenson JM, Lim S, Fraser SDS, Roberts HC. A systematic review of the evidence for deprescribing interventions among older people living with frailty. BMC Geriatr. 2021 Apr 17;21(1):258. doi: 10.1186/s12877-021-02208-8. PMID 33865310
- [Background] Pazan F, Wehling M. Polypharmacy in older adults: a narrative review of definitions, epidemiology and consequences. Eur Geriatr Med. 2021 Jun;12(3):443-452. doi: 10.1007/s41999-021-00479-3. Epub 2021 Mar 10. PMID 33694123